CLINICAL TRIAL: NCT03217968
Title: Abortive Treatment of Migraine With the Cefaly® Abortive Program Device: Pilot Trial
Brief Title: Abortive Treatment of Migraine With the Cefaly® Abortive Program Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50803
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Results first posted 2018-06-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active (Experimental): 120 minutes of Cefaly® Abortive Program device stimulation as abortive treatment of an early stage migraine attack
  Interventions: Device: Cefaly® Abortive Program device

INTERVENTIONS:
Device: Cefaly® Abortive Program device — The Cefaly® Abortive Program device is an external cranial neurostimulator designed for supraorbital neurostimulation, also known as external Trigeminal Nerve Stimulation (e-TNS).

SUMMARY:
The purpose of this study is to investigate the efficacy of the Cefaly® Abortive Program device used at home for 2 hours to treat a migraine attack. This open clinical trial will study the abortive treatment of migraine using the Cefaly® Abortive Program device, prior to development of a sham-controlled trial.

DETAILED DESCRIPTION:
The main objective of this study is to have a pilot assessment of the efficacy of the Cefaly® Abortive Program device used at home for 2 hours to treat a migraine attack, as triptans are generally used. That is to say having pilot data to assess the efficacy of the Cefaly® Abortive Program device in the abortive treatment of acute migraine as measured by 2-hour pain freedom, pain relief and migraine associated symptoms freedom, plus evolution of these measurements for 24 hours after the beginning of the treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years on the day of signing the informed consent form
* ≥ 1-year history of migraine with or without aura according to the diagnostic criteria listed in the International Classification of Headache Disorders (ICHD)-III beta (2013) section 1, migraine (8), with the exception of aura without headache, hemiplegic migraine and brainstem aura migraine
* Migraine onset before the age of 50 years
* Having between 2 and 8 moderate or severe migraine attacks (Grade 2 or 3) per month in each of the two months prior to screening
* Patient understands the study procedures, alternative treatments available, and voluntarily agrees to participate in the study by giving written informed consent
* Patient is able to read and understand the written information (instruction sheet, paper diary and Adverse Events (AE) collecting form)

Exclusion Criteria:

* Patient has difficulty distinguishing his/her migraine attacks from tension-type headaches
* Patient has more than 15 headache days per month
* Patient having received supraorbital nerve blocks in the prior 4 months
* Patient having received Botox treatment in the prior 4 months
* Modification of a migraine prophylaxis treatment in the previous 3 months
* Diagnosis of other primary headache disorders, except rare (< 4) tension-type headaches per month
* Diagnosis of secondary headache disorders included Medication Overuse Headache
* Patients abusing opioids or user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence
* Implanted metallic or electronic device in the head
* Cardiac pacemaker or implanted or wearable defibrillator
* Patient having had a previous experience with the Cefaly® device
* Migraine Aura without headache
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of screening visit (Visit 1)
* Patients not having the ability to use appropriately the device and/or to perform themselves or bear the first 20-minute stimulation session during the training session at the study site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph MANN, M.D., Principal Investigator — Rochester Clinical Research
Locations (1):
- Rochester Clinical Research, Inc., Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active
Started | 59
Completed | 48
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Arm/Group | Active
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.85 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Migraine type [Count of Participants; unit: Participants]
  Migraine with aura | 15
  Migraine without aura | 33
Migraine intensity [Count of Participants; unit: Participants]
  Moderate intensity at baseline | 33
  Severe intensity at baseline | 15
Most bothersome syndrome [Count of Participants; unit: Participants]
  Nausea | 11
  Vomiting | 1
  Sensitivity to light | 27
  Sensitivity to sound | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain Freedom (PF) at 2 Hours
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to no headache (Grade 0) at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 17

2. Primary Outcome: Most Bothersome Migraine-associated Symptom (MBS) Freedom at 2 Hours
Description: The percentage of patients with absence, at 2 hours after the beginning of the e-TNS session, of the most bothersome migraine-associated symptom identified at baseline.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 29

3. Secondary Outcome: Pain Relief (PR) at 2 Hours
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 34

4. Secondary Outcome: Migraine-associated Symptoms Freedom at 2 Hours
Description: The percentage of patients with absence of photophobia, phonophobia, nausea and vomiting, at 2 hours after the beginning of the e-TNS session.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 22

5. Secondary Outcome: Use of Rescue Medication Between 2 and 24 Hours
Description: The percentage of patients who took acute anti-migraine medication between 2 and 24 hours after the beginning of the e-TNS session.
Time Frame: Between 2 and 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 24

6. Secondary Outcome: Sustained Pain Freedom at 24 Hours
Description: The percentage of patients having no headache (Grade 0) at 2 hours, with no use of rescue medication and no relapse of headache pain within the 24 hours after the beginning of the e-TNS session.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 48
Participants | 12

ADVERSE EVENTS:
Time Frame: The data was collected during the 24 hours following the start of the treatment
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 15/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=59)
Burning sensation on the forehead (Skin and subcutaneous tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 1 (1)
itching/tingling/stinging/numbness sensation on forehead (Skin and subcutaneous tissue disorders) | 4 (4)
Nausea (Nervous system disorders) | 2 (2)
Vomiting (Nervous system disorders) | 1 (1)
Pain in the jaw (Nervous system disorders) | 1 (1)
Discomfort in teeth (Nervous system disorders) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1)
Cold feet (Blood and lymphatic system disorders) | 1 (1)
Pain in eyes (Nervous system disorders) | 1 (1) — Severe pain in eyes when eyes open while wearing device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 90 days from the time submitted to the sponsor for review. Sponsor may request:

* deletion of any trade secret, proprietary, or confidential information of Sponsor
* an additional 90 days to take measures to preserve its Intellectual Property rights

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03217968/Prot_SAP_000.pdf